CLINICAL TRIAL: NCT06392750
Title: PWP1 Affects Gastric Cancer Progression by Regulating p53 and JAK1 and Its Expression in Gastric Cancer.
Brief Title: PWP1's Expression in Gastric Cancer.
Status: Completed | Type: Observational
Sponsor: Northern Jiangsu People's Hospital (Other)
Responsible Party: Principal Investigator, Daorong Wang, Professor, M.D., Northern Jiangsu People's Hospital
Other Study IDs: mj2404001
Record Dates: First submitted 2024-04-26; First posted 2024-04-30 (Actual); Last update posted 2024-04-30 (Actual); Status verified 2024-04

CONDITIONS: Diagnosis; Gastric Cancer
Keywords: gastric cancer; PWP1; IHC; expression
MeSH Terms: conditions — Disease; Stomach Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples Without DNA — Apply to the biological sample library for samples of tumor tissue and adjacent tissues preserved during surgery in gastric cancer patients. Subsequently, prepare tissue slices for immunohistochemical staining and compare the expression profiles between the two sample groups.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- adjacent tissues: Paraffin tissue microarray slides prepared from normal tissue adjacent to tumor tissue removed during gastrectomy were retrieved from the biological sample library of the Northern Jiangsu People's Hospital.
- tumor tissues: Paraffin tissue microarray slides prepared from tumor tissue removed during gastrectomy were retrieved from the biological sample library of the Northern Jiangsu People's Hospital.
  Interventions: Behavioral: Collection of tumor tissue specimens

INTERVENTIONS:
Behavioral: Collection of tumor tissue specimens — Collection of tumor tissue specimens during surgery
  Groups: tumor tissues

SUMMARY:
Background：Gastric cancer is a globally important disease and the fifth most diagnosed malignant cancer in the world. Because it is usually diagnosed at an advanced stage, gastric cancer has a high mortality rate, making it the third most common cause of cancer-related death. Hot spots of gastric cancer incidence and mortality exist in East Asia, Eastern Europe and South America. It is still an urgent problem to find new diagnostic and prognostic markers and better understand the molecular mechanism of gastric cancer. Although radical resection and systemic chemotherapy have shown great improvement, the prognosis of gastric cancer (GC) patients is still depressing due to malignant proliferation and metastasis. Therefore, it is urgent to clarify the potential molecular mechanism of gastric cancer progression, which will contribute to the development of targeted therapy. Effective induction of tumor cell apoptosis is the most important feature of a new chemical agent for cancer treatment. There is increasing evidence that the cell cycle can act in concert with apoptosis to cause cell death under certain cellular stress conditions. A comprehensive understanding of the relationship between apoptosis and cell cycle is essential for developing effective cancer therapies.

PWP1 is also known as endonuclein, which contains five WD40 repeated domains and belongs to the WD40-repeated superfamily. It is highly expressed in human pancreatic adenocarcinoma, where it functions as a cell-cycle regulator. However, the normal function of Pwp1 is largely unknown. Previous research data show that PWP1 plays a key role in regulating biological functions such as RNA processing, signal transduction, gene expression, vesicle transport, cytoskeleton assembly and cell cycle progression. Whether the high expression of PWP1 is ubiquitous in tumors, the relationship between the high expression and clinicopathological factors of tumors, and the mechanism of PWP1 in tumors are still unclear. Further exploration of the molecular mechanism of PWP1 in GC may provide new ideas and therapeutic targets for GC treatment in the future, and benefit clinical patients.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed as gastric cancer
* Performing gastric cancer resection surgery
* Informed consent signed prior to surgery.

Exclusion Criteria:

* Emergency surgery
* Preoperative and intraoperative detection of distant organ metastases or extensive
* No standard chemotherapy for tumor-node-metastasis (TNM) staging II or III after surgery
* Incomplete case data.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: A total of 200 gastric cancer patients, including 80 (40.0%) men and 120(60.0%) women, were enrolled in this study.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2021-05-01 (Actual); Primary Completion 2023-10-30 (Actual); Study Completion 2024-04-01 (Actual)

PRIMARY OUTCOMES:
The expression of PWP1 in adjacent tissues and tumor tissues of patients with gastrectomy for gastric cancer. | 6 to 12 months after operation
  Test the expression of PWP1 in adjacent tissues and tumor tissues of patients with gastrectomy for gastric cancer through the immunohistochemical.

CONTACTS AND LOCATIONS:
Overall Officials: Daorong Wang, M.D., Professor, Study Director — Northern Jiangsu People's Hospital
Locations (1):
- Northern Jiangsu People's Hospital Affiliated to Yangzhou University, General Surgery Institute of Yangzhou, Yangzhou University , Yangzhou, Yangzhou, Jiangsu, China

IPD SHARING:
Plan to Share IPD: Undecided
Contains a large amount of personal information about patients and needs to be treated with caution.